CLINICAL TRIAL: NCT03372434
Title: Clinical Investigation of the TECNIS Next-Generation Intraocular Lens
Brief Title: Clinical Investigation of the Next-Generation Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUR-CAT-652-1001
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Investigational Lens Device #1 (Experimental): Investigational Intraocular Lens Device #1: Model ZFR00
  Interventions: Device: Investigational Intraocular Lens Device #1: Model ZFR00
- Investigational Lens Device #2 (Experimental): Investigational Intraocular Lens Device #1: Model ZYR00
  Interventions: Device: Investigational Intraocular Lens Device #1: Model ZYR00
- Control Device (Active Comparator): Control TECNIS Multifocal Intraocular Lens Model ZLB00
  Interventions: Device: TECNIS Multifocal Intraocular Lens: Model ZLB00

INTERVENTIONS:
Device: Investigational Intraocular Lens Device #1: Model ZFR00 — IOL replaces the natural lens removed during cataract surgery.
  Arms: Investigational Lens Device #1
Device: Investigational Intraocular Lens Device #1: Model ZYR00 — IOL replaces the natural lens removed during cataract surgery.
  Arms: Investigational Lens Device #2
Device: TECNIS Multifocal Intraocular Lens: Model ZLB00 — IOL replaces the natural lens removed during cataract surgery.
  Arms: Control Device

SUMMARY:
This study is a 6-month, prospective, multicenter, subject/evaluator-masked, bilateral, randomized clinical investigation of the TECNIS Next-Generation Model ZFR00 and Model ZYR00 IOLs versus the TECNIS Multifocal Model ZLB00 control IOL.

The study will be conducted at up to 14 sites in the U.S.A and will enroll up to 260 subjects to achieve approximately 220 randomized and bilaterally-implanted subjects, resulting in approximately 195 evaluable subjects (65 in each test group and 65 in the control group) at 1 and 6 months. Subjects are to be implanted with the same IOL in both eyes, the ZFR00 IOL, the ZYR00 IOL or the ZLB00 control IOL. The eye implanted first will be considered the primary study eye.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age
* Bilateral cataracts for which posterior chamber IOL implantation has been planned
* Preoperative best corrected distance visual acuity (BCDVA) of 20/40 Snellen or worse with a glare source or 20/40 Snellen or worse without a glare source
* Potential for postoperative BCDVA of 20/30 Snellen or better
* Corneal astigmatism:

  * Normal corneal topography
  * Preoperative corneal astigmatism of 1.00 D or less in both eyes
* Clear intraocular media other than cataract in each eye
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries
* Ability to understand and respond to a questionnaire in English

Exclusion Criteria:

* Requiring an intraocular lens power outside the available range of +14.0 D to +26.0 D
* Any clinically-significant pupil abnormalities (non-reactive, fixed pupils, or abnormally-shaped pupils)
* Irregular corneal astigmatism
* Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
* Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery. Note: Prophylactic peripheral iridotomies and peripheral laser retinal repairs that, in the opinion of the investigator will not confound study outcome or increase risk to the subject, are acceptable.
* Corneal abnormalities such as stromal, epithelial or endothelial dystrophies that are predicted to cause visual acuity losses to a level worse than 20/30 Snellen during the study
* Inability to achieve keratometric stability for contact lens wearers (per procedure outlined in Section 10.3)
* Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
* Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause visual acuity losses to a level worse than 20/30 Snellen during the study
* Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects
* Use of systemic or ocular medications that may affect vision
* Prior, current, or anticipated use during the course of the 6-month study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) that may, in the opinion of the investigator, confound the outcome or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery)
* Poorly-controlled diabetes
* Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.). Note: controlled ocular hypertension without glaucomatous changes (optic nerve cupping and visual field loss) is acceptable.
* Known ocular disease or pathology that, in the opinion of the investigator,

  * may affect visual acuity
  * may require surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, uncontrolled glaucoma, etc.)
  * may be expected to require retinal laser treatment or other surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, etc.)
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
* Concurrent participation or participation within 60 days prior to preoperative visit in any other clinical trial
* Desire for monovision correction

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbott Medical Optics Clinical Trials, Study Director — Abbott Medical Optics
Locations (12):
- United States (12):
  - Empire Eye & Laser Center, Bakersfield, California
  - Katzen Eye Care and Laser Center, Boynton Beach, Florida
  - Chesapeake Eye Care & Laser Center, Annapolis, Maryland
  - Eye Doctors of Washington, Chevy Chase, Maryland
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Carolina EyeCare Physicians, LLC, Mt. Pleasant, South Carolina
  - Loden Vision Centers, Goodlettsville, Tennessee
  - Eye Specialty Group, Memphis, Tennessee
  - Texas Eye and Laser Center, Hurst, Texas
  - Lehmann Eye Center, Nacogdoches, Texas
  - Focal Point Vision, San Antonio, Texas
  - Clarus Eye Centre, Lacey, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 225 subjects were implanted with a study lens in at least one eye. Two hundred and twenty five (225) subjects had a study IOL in the first eye.
Units Other Than Participants: Eyes
Groups:
- Model ZFR00; Model ZYR00: Investigational IOL implanted in the first eye
- Model ZLB00: Control IOL implanted in the first eye
Period: Overall Study
Arm/Group | Model ZFR00 | Model ZLB00 | Model ZYR00
Started (Implanted with a study lens in at least one eye) | 78; 78 Eyes | 73; 73 Eyes | 74; 74 Eyes
1 Month Follow-up | 76; 76 Eyes | 72; 72 Eyes | 73; 73 Eyes
Completed (6 months follow up) | 76; 76 Eyes | 70; 70 Eyes | 72; 72 Eyes
Not Completed | 2; 2 Eyes | 3; 3 Eyes | 2; 2 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Model ZFR00 | Model ZLB00 | Model ZYR00 | Total
Number analyzed (Participants) | 78 | 73 | 74 | 225
Age, Customized [Number; unit: Participants]
  Less than <60 years | 10 | 13 | 17 | 40
  60-69 years | 38 | 35 | 34 | 107
  70-79 years | 27 | 23 | 21 | 71
  Greater than or equal to >/80 years | 3 | 2 | 2 | 7
  Not reported | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 48 | 49 | 151
  Male | 24 | 25 | 25 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 3 | 13
  Not Hispanic or Latino | 74 | 67 | 71 | 212
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (including Indian) | 0 | 3 | 0 | 3
  Black | 3 | 7 | 7 | 17
  Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0
  Caucasian | 75 | 62 | 66 | 203
  Another Race | 0 | 1 | 0 | 1
  Not reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Distance Corrected Intermediate Visual Acuity
Description: Visual Acuity (VA) was assessed monocularly (each eye separately) under photopic (well-lit) conditions using best distance correction (distance refraction) and high contrast, Early Treatment Diabetic Retinopathy Study (ETDRS) chart at 66 cm from spectacle plane. It was measured in logarithm of the minimum angle of resolution (logMAR), on an ETDRS chart. A lower numeric value represented better VA. This analysis was pre-specified for the first operative eye only.
Time Frame: 1 month
Population: Safety population
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Model ZFR00 | Model ZLB00 | Model ZYR00
Number analyzed (Participants) | 76 | 72 | 73
Number analyzed (Eyes) | 76 | 72 | 73
LogMAR | 0.098 (0.115) | 0.219 (0.146) | 0.147 (0.149)

ADVERSE EVENTS:
Time Frame: 6 months
Description: All Serious Adverse Events (device related and non-device related) are reported. Device related non-serious adverse events are reported as Other Adverse Events.
Groups:
- Model ZFR00; Model ZYR00: Investigational IOL device
- Model ZLB00: Control IOL Device
Arm/Group | Model ZFR00 | Model ZLB00 | Model ZYR00
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/73 | 0/74
Serious Adverse Events (participants affected / at risk) | 5/78 | 13/73 | 4/74
Other Adverse Events (participants affected / at risk) | 6/78 | 1/73 | 3/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model ZFR00 (N=78) | Model ZLB00 (N=73) | Model ZYR00 (N=74)
Cystoid Macular Edema (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Macular Hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Bothersome Visual Symptom (Product Issues) | 1 (1) | 1 (1) | 1 (1) — Adverse Device Effect due to report of bothersome visual symptoms causing significant impairment lasting more than 3 months postoperatively
Herpes Zoster Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual symptoms requiring secondary surgical intervention (Product Issues) | 1 (1) | 0 (0) | 1 (1)
Haptic anterior to capsule bag (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Increase in cells likely due to non-compliance with ocular medication regimen (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal Hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Hospitalization (General disorders) | 0 (0) | 3 (3) | 1 (1)
Patent Foramen Ovale (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angioplasty (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
B-cell Lymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — with permanent nerve damage
Undisclosed illness requiring Hospice care (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model ZFR00 (N=78) | Model ZLB00 (N=73) | Model ZYR00 (N=74)
Bothersome visual symptom (Product Issues) | 6 (6) | 1 (1) | 3 (3) — Adverse Device Effect due to report of bothersome visual symptoms causing significant impairment lasting more than 3 months postoperatively

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at anytime

DOCUMENTS (2):
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03372434/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT03372434/SAP_001.pdf